CLINICAL TRIAL: NCT06055621
Title: Evaluation of DASATINIB Monotherapy in Acute Myeloid Leukemia Patients Refractory to VENETOCLAX-AZACITIDINE
Brief Title: Evaluation of DASATINIB Monotherapy Efficacy in Acute Myeloid Leukemia Patients Refractory to VENETOCLAX-AZACITIDINE
Acronym: VEN-R DASA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEN-R DASA-IPC 2022-067
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DASATINIB (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Daily orally administration of DASATINIB

SUMMARY:
The goal of this clinical trial is to learn about the efficacy of DASATINIB monotherapy in acute myeloid leukemia patients refractory to VENETOCLAX-AZACITIDINE. The main question it aims to answer is to assess the tumor response after 2 cycles of DASATINIB monotherapy treatment for patients with chemotherapy-ineligible acute myeloid leukemia refractory to VENETOCLAX-AZACITIDINE therapy.

Participants will be given DASATINIB treatment up to 3 months. Response will be assessed by a myelogram and a complete blood count at the end of every cycle. Follow up will last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML except Philadelphia chromosome-positive AML (Ph+) and acute promyelocytic leukemia (AML M3)
* Age ≥ 18 years
* ECOG ≤3
* VEN-AZA refractory defined as no response after two cycles of VEN-AZA whatever the dose and the treatment duration
* Signed informed consent form
* Affiliation to a social security system, or beneficiary of such a system

Exclusion Criteria:

* Patient eligible to a targeted therapy having a market authorization
* Central nervous system involvement
* Heart failure
* Liver failure
* Kidney failure
* Contraindication to DASATINIB
* Positive for HIV (detectable viral load), Hepatitis B or C
* Pregnant or breastfeeding woman
* No efficient contraception for the women of childbearing age
* Emergency situation person or not able to express his/her informed consent
* Patient under a legal protection measure (adult under guardianship, curatorship or safeguard of justice)
* Inability to undergo the clinical trial medical follow-up for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
tumor response | 2 months
  Objective response rate after 2 cycles of 28 days DASATINIB defined as the rate of complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) according to ELN 2022 criteria.

SECONDARY OUTCOMES:
response rates | 3 months
  Different response rates (RC, CRi, or partial remission (PR)) according to ELN 2022 criteria.
Time to response | 3 months
  Time to response (time between the start of the treatment until achievement of the CR, CRi or PR)
Duration of relapse-free period | 3 months
  Duration of relapse-free period (time between the response time and the relapse)
Event-free survival | 3 months
  Event-free survival (EFS, time between start of treatment and relapse, no response or death)
Overall survival | 3 months
  Overall survival (duration of survival from the start of the treatment)
Occurrence of Adverse Events | 3 months
  Occurrence of Adverse Events according to CTCAE v5.0 and Serious Adverse Reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No